CLINICAL TRIAL: NCT05314309
Title: Clinical Validation of a Multi-target Faecal Immunochemical Test (mtFIT) Versus a Faecal Immunochemical Test (FIT) for Detecting Advanced Neoplasia in Population Screening for CRC: a Prospective Cohort Study With Paired Design
Brief Title: Prospective Clinical Validation of a Novel Multitarget FIT in CRC Screening
Acronym: mtFIT
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: The Netherlands Cancer Institute (Other)
Collaborators: Amsterdam University Medical Centers (UMC), Location Academic Medical Center (AMC) (Other); Erasmus Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: M22ANC; 1691110-204907-PG (Other: Dutch Ministry of Health, Welfare and Sport (VWS))
Record Dates: First submitted 2022-02-14; First posted 2022-04-06 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2023-01

CONDITIONS: CRC; Advanced Neoplasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- mtFIT: Individuals who consent to participate in the study, will be asked to take two stool samples from the same bowel movement. In a central laboratory these two samples then will be analyzed. One with the standard of care faecal immunochemical test (FIT) and the other with the multi-target faecal immunochemical test (mtFIT). If either one of these two tests is positive, individuals will be referred to undergo a colonoscopy procedure. The performance of mtFIT, in comparison to FIT, will be evaluated against the colonoscopy findings.
  Interventions: Diagnostic Test: Comparison of two tests (FIT and mtFIT) in the same bowel movement

INTERVENTIONS:
Diagnostic Test: Comparison of two tests (FIT and mtFIT) in the same bowel movement — Invitees for the Dutch National CRC screening program will be randomly selected by the Screening Organization and invited to participate in this study, where next to the current FIT, participants will also perform the mtFIT in one bowel movement. Both tests will be analysed and if one of the two test results is positive, the individual will be referred for colonoscopy.

SUMMARY:
The primary goal of the population-based colorectal (CRC) screening is early detection and interception of CRC and its precursors to decrease CRC-related morbidity and mortality. To improve current CRC screening programs, the investigators have developed and retrospectively validated a test that combines the detection of multiple proteins in stool (the multitarget faecal immunochemical test, mtFIT). mtFIT was found to have a higher accuracy to detect advanced neoplasia (AN), which includes CRC, advanced adenomas and advanced serrated polyps, in comparison to FIT. Thus, this multitarget test has the potential to improve the screening program's efficiency in reducing CRC-related incidence, morbidity and mortality. This new test, in comparison to FIT, shows specifically higher sensitivity in the detection of advanced adenomas, without affecting specificity.

DETAILED DESCRIPTION:
Background:

The primary goal of population-based CRC screening is early detection and interception of CRC and its precursors to decrease CRC-related morbidity and mortality. New tests, with higher sensitivity for advanced precursor lesions than the current FIT, are desired. The investigators have developed a protein-based multitarget faecal immunochemical test (mtFIT) that shows higher sensitivity for advanced adenomas without losing in specificity.

Objective:

To prospectively validate the better performance of the mtFIT in comparison to FIT in the setting of a population-based CRC screening program.

Material and Methods:

In this prospective study, participants of the Dutch National CRC screening program (55-75 years of age) will be invited to participate. Individuals who consent to participate in the study, will be asked to take two stool samples from the same bowel movement. In a central laboratory these two samples then will be analyzed. One with the standard of care faecal immunochemical test (FIT) and the other with the multi-target faecal immunochemical test (mtFIT). If either one of these two tests is positive, individuals will be referred to undergo a colonoscopy procedure. The performance of mtFIT, in comparison to FIT, will be evaluated against the colonoscopy findings.

Expected results:

mtFIT has higher sensitivity for AN, and in particular advanced adenomas, than FIT, at equal positivity rate.

ELIGIBILITY:
Inclusion Criteria:

* Individuals of the Dutch population suitable for CRC screening (age between 55 and 75 years old) will be randomly selected.
* The participants will be invited in phases and are selected out of different age groups.
* The selected participants will participate in the population CRC screening program for either the first, second, third or fourth time.

Exclusion Criteria:

* Collection of stool not complete for both tests (FIT and mtFIT)

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The intended population of this study consists of subjects participating in the national Dutch National CRC screening program
Sampling Method: Non-Probability Sample
Enrollment: 14712 (Actual)
Dates: Start 2022-03-25 (Actual); Primary Completion 2023-05-31 (Estimated); Study Completion 2023-05-31 (Estimated)

PRIMARY OUTCOMES:
Detection rate of advanced neoplasia | 10 months
  Relative sensitivity of mtFIT compared to FIT in the detection of advanced neoplasia (AN; CRC, advanced adenomas and advanced serrated polyps) at an equal positivity rate.

SECONDARY OUTCOMES:
Diagnostic yield of mtFIT in comparison to FIT | 10 months
  mtFIT detects more CRC, more early-stage CRC and more advanced polyps (advanced adenomas and advanced serrated polyps) compared to FIT.

OTHER OUTCOMES:
Long-term mtFIT efficacy | 10 months
  mtFIT reduces CRC incidence and CRC-related mortality compared to FIT and is cost-effective to be used in a CRC screening program.

CONTACTS AND LOCATIONS:
Overall Officials: Gerrit A Meijer, MD, PhD, Principal Investigator — The Netherlands Cancer Institute; Evelien Dekker, MD, PhD, Study Chair — Amsterdam University Medical Centers (UMC), Location Academic Medical Center (AMC); Manon CW Spaander, MD, PhD, Study Chair — Erasmus University Medical Centre Rotterdam (Erasmus MC)
Locations (1):
- Netherlands Cancer Institute, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wisse PHA, de Klaver W, van Wifferen F, van Maaren-Meijer FG, van Ingen HE, Meiqari L, Huitink I, Bierkens M, Lemmens M, Greuter MJE, van Leerdam ME, Spaander MCW, Dekker E, Coupe VMH, Carvalho B, de Wit M, Meijer GA. The multitarget faecal immunochemical test for improving stool-based colorectal cancer screening programmes: a Dutch population-based, paired-design, intervention study. Lancet Oncol. 2024 Mar;25(3):326-337. doi: 10.1016/S1470-2045(23)00651-4. Epub 2024 Feb 9. PMID 38346438
- [Derived] Wisse PHA, de Klaver W, van Wifferen F, Meiqari L, Bierkens M, Greuter MJE, Carvalho B, van Leerdam ME, Spaander MCW, Dekker E, Coupe VMH, de Wit M, Meijer GA. The multitarget fecal immunochemical test versus the fecal immunochemical test for programmatic colorectal cancer screening: a cross-sectional intervention study with paired design. BMC Cancer. 2022 Dec 12;22(1):1299. doi: 10.1186/s12885-022-10372-2. PMID 36503495